CLINICAL TRIAL: NCT05922917
Title: Pulmonary Vein Isolation Versus Complex Procedure Using Pulsed-field Ablation in Patients With Persistent Atrial Fibrillation
Brief Title: Pulsed-field Ablation in Patients With Persistent Atrial Fibrillation
Acronym: PIVCO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: České Budějovice Hospital (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZ-060620231904
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Persistent Atrial Fibrillation; Pulsed-field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI (Active Comparator): Pulmonary vein isolation
  Interventions: Device: pulsed-field ablation
- PVI+ (Experimental): Pulmonary vein isolation supplemented by the additional lesions: left atrial posterior wall isolation, mitral and cavotricuspid isthmus lines
  Interventions: Device: pulsed-field ablation

INTERVENTIONS:
Device: pulsed-field ablation — application of pulsed-field energy for pulmonary vein isolation and linear ablations

SUMMARY:
Since a new method called pulsed-field ablation (PFA) has emerged, allowing significantly simpler, safer, and faster creation of ablative lesions in paroxysmal AF and PsAF (13), redefining the "optimal" ablation approach started to appear mandatory. Our project (The PIVCO study) aims to determine a more standardized procedure representing optimal ablation strategy for patients suffering from PsAF using PFA and multielectrode ablation catheters. The central hypothesis is that ablation of the posterior LA wall (PWI), together with mitral and cavotricuspid isthmus ablation added on top of PVI, will be associated with better effects in terms of rhythm control. Given the speed, safety, and ease of standardization of ablation using electroporation, a demonstration of the superiority of either approach could significantly impact the current standard of clinical care.

DETAILED DESCRIPTION:
Purpose Since a new method called pulsed-field ablation (PFA) has emerged, allowing significantly simpler, safer, and faster creation of ablative lesions in paroxysmal AF and PsAF (13), redefining the "optimal" ablation approach started to appear mandatory. Our project (The PIVCO study) aims to determine a more standardized procedure representing optimal ablation strategy for patients suffering from PsAF using PFA and multielectrode ablation catheters. The central hypothesis is that ablation of the posterior LA wall (PWI), together with mitral and cavotricuspid isthmus ablation added on top of PVI, will be associated with better effects in terms of rhythm control. Given the speed, safety, and ease of standardization of ablation using electroporation, a demonstration of the superiority of either approach could significantly impact the current standard of clinical care.

Primary endpoints

(1) The primary endpoint will be a recurrence of AF (or atrial tachycardia, AT) lasting >30 seconds as assessed using repeated 7-day ECG Holter monitoring in patients without anti-arrhythmic drugs (AADs) during the entire post-blanking follow-up, i.e., starting three months after the index procedure. All patients should complete a 12-month follow-up period.

Secondary endpoints

(1) The first recurrence of on-AADs AF/AT lasting >6 minutes during the post-blanking follow-up period (i.e., disregarding all off-AAD episodes). (2) Number of hospitalizations and emergency out-patient visits related to AF/AT recurrence, worsening of heart failure, or other cardiovascular diseases. (3) Number of electrical cardioversions. (4) Proportion of patients on AADs at the end of follow-up. (5) PFA-related complications. (6) Assessment of the quality of life using standardized instruments (AFEQT, EQ5D). (7) Feasibility of achieving a complete block of the mitral isthmus and PWI using PFA (8) Proportion of patients with delayed conduction into LAA after mitral line (9) Number of patients that underwent repeated ablations during follow-up.

Interventions

Procedures that will be performed on the day of admission for ablation:

1. 12-lead ECG
2. Randomization to group PVI or PVI+
3. Physical examination
4. Medication taken
5. Medical history
6. Laboratory tests (biochemistry - NTproBNP, K, urea, creatinine, ALT, AST, GMT, CRP; KO - Hb, leu, PLT)
7. Cardiac CT scan as decided by the attending physician
8. Transthoracic echocardiography (left atrial [LA] dimension in PLAX, LAVi, transverse and longitudinal LA dimension in A4CH, LA area in A4CH, left ventricular ejection fraction (LV EF), LV dimension in PLAX, estimation of PASP, quantification of any valvular defect
9. Esophageal echocardiography (TEE) of the heart as decided by the attending physician to exclude intracardiac thrombosis
10. Quality of life questionnaires (EQ5DY, AFEQT)

Catheter ablation strategy

In all patients, ablation will be performed by electroporation (Farapulse system), as recommended, with at least two applications per each ablation spot. Based on the randomization, patients will be treated using two distinct approaches:

Group PVI (Pulmonary vein isolation only)

1. No ablation at the cavotricuspid isthmus (CTI)
2. Transseptal puncture
3. PVI (plus application to the superior anterior aspect of the right superior pulmonary vein [RSPV])
4. In the absence of AF termination - cardioversion
5. Induction - in case of persistent arrhythmia (regardless of regularity of activation in the atria) - cardioversion, without further ablation outside PVI

Group PVI+ (Complex ablation procedure)

1. Transseptal puncture
2. PVI (plus application to the superior anterior aspect of the RSPV)
3. Roofline
4. Box isolation of the posterior wall of the left atrium (line on the LA roof between left superior pulmonary vein [LSPV] and RSPV, the line between left inferior pulmonary vein [LIPV] and right inferior pulmonary vein [RIPV])
5. Ablation along the coronary sinus (CS) from the endocardium, in the form of limited energy application in the left postero-septum
6. Posterolateral mitral isthmus line
7. In the absence of termination of AF to SR or when AF is converted to AT, cardioversion will be performed
8. Verification and eventual completion of the bidirectional mitral line conduction block
9. Ablation at CTI - completion of the bidirectional conduction block
10. Induction (burst atrial pacing from proximal CS at different cycle lengths of 300 ms, 250 ms, and 200 ms, each step for 5-10 seconds; then RAMP pacing 300-200 ms)
11. If AF or AT is induced, cardioversion will be performed

Follow-up The following information will be recorded on the day of discharge: Date of hospital discharge after ablation, length of in-hospital stays, early complications of ablation, and medication at the discharge (all antiarrhythmic drugs except beta-blockers will permanently be discontinued at hospital discharge).

Four 7-day Holter ECG monitoring recordings will be done at 3, 6, 9, and 12 months after ablation (in case of recurrence of AF after ablation, standard treatment according to the treating physician's decision, including the possibility of antiarrhythmic medication, electrical cardioversion or repeated ablation, will be applied).

A telephone visit be done at 1, 3, 6, and 9 months after ablation with an inquiry about complications of the ablation procedure, perceived recurrence of AF, use of antiarrhythmic and antithrombotic medication, elective cardioversion, hospitalization, and reasons for it.

An in-office visit will be done 12 months after ablation in the hospital's out-patient department, including an inquiry about complications of the ablation procedure, perceived and documented recurrence of AF, use of antiarrhythmic and antithrombotic medication, elective cardioversion, hospitalization and reasons for it after ablation, physical examination, medication history, ECG, echocardiography and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or long-standing persistent AF proved on at least two 12-lead ECG recordings more than one week apart or > 7-day EKG Holter recordings
* Age ≥ 18 years at the time of study enrollment
* Signed informed consent

Exclusion Criteria:

* Paroxysmal AF
* Sinus rhythm on the 12-lead ECG on admission unless recent external electrical cardioversion was carried out within the last six months and the patient is treated by amiodarone
* LA diameter > 55 mm (measured in the parasternal long-axis view)
* History of AF ablation in the past
* History of cardiac surgery
* Significant valvular defect
* Age below 18 years
* Pregnancy, breastfeeding
* Any disease with a life expectancy <1 year
* Terminal renal failure
* History of pacemaker or defibrillator implantation
* Significant thyroid disease
* Uncorrected congenital heart disease or valvular obstruction
* Obstructive hypertrophic cardiomyopathy
* Active myocarditis
* Constrictive pericarditis
* Untreated hypothyroidism or hyperthyroidism
* Adrenal insufficiency
* Active vasculitis due to collagen vascular disease
* Presence on a heart transplant waiting list (UNOS category 1A or 1B or equivalent). Patients on a non-acute heart transplant waiting list (UNOS category 2 or 7 or equal) are eligible for inclusion in the study
* Recipient of any major organ transplant (e.g., lung, liver, heart)
* Patient who is undergoing or has undergone cytotoxic or cytostatic chemotherapy and radiation therapy for the treatment of malignancy within six months before randomization or clinical evidence of current malignancy, with the following exceptions: basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, prostate cancer (if the localized disease is stable, with life expectancy > 2.5 years in the opinion of the investigator)
* HIV positivity with a survival expectancy of less than five years due to HIV
* Chronic kidney disease with glomerular filtration rate < 30 ml/min
* Chronic dialysis treatment
* Recent (within three months) self-reported history of alcoholism or illicit drug dependence
* Any illness (e.g., psychiatric illness) or situation that, in the opinion of the investigator, could place the subject at significant risk, confound the results of the study, or significantly affect the subject's participation in the study
* Unwillingness to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 1 year following ablation procedure
  The primary endpoint will be a recurrence of AF (or atrial tachycardia, AT) lasting >30 seconds as assessed using repeated 7-day ECG Holter monitoring in patients without anti-arrhythmic drugs (AADs) during the entire post-blanking follow-up, i.e., starting three months after the index procedure. All patients should complete a 12-month follow-up period.

SECONDARY OUTCOMES:
Atrial fibrillation recurrence on AADs | 1 year following ablation procedure
  The first recurrence of on-AADs AF/AT lasting >6 minutes during the post-blanking follow-up period (i.e., disregarding all off-AAD episodes).
Hospitalization rate | 1 year following ablation procedure
  Number of hospitalizations and emergency out-patient visits related to AF/AT recurrence, worsening of heart failure, or other cardiovascular diseases.
Cardioversion | 1 year following ablation procedure
  Number of electrical cardioversions.
Complications | 1 year following ablation procedure
  PFA-related complications.
Atrial Fibrillation Effect on Quality of Life (AFEQT) | 1 year following ablation procedure
  Assessment of the quality of life using standardised instrument AFEQT. Three domains and global QoL will be assessed using a calculated score of 0 to 100% (100% = the best quality of life) based on the patient´s response to 20 questions.
EuroQol Group questionnaire on quality of life | 1 year following ablation procedure
  Assessment of mobility, self-care, pain or discomfort, anxiety or depression by a Likert scale (1-3, 1 = no limitation, 3 = severe limitation) complemented by visual aid score (1-100, the higher score, the better quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Ceske Budejovice Hospital, České Budějovice, Czechia

IPD SHARING:
Plan to Share IPD: No